# Official Title of the study: Effects of Altered Auditory Feedback on Speech Fluency

**NCT Number:** [NCT ID not yet assigned]

**Date:** 05/01/2023

# **Study Details:**

The Mumble Melody Longitudinal Study is a month long online study in which we will be investigating the longer term effects of using the Mumble Melody app for people who stutter. During the course of a month, eligible participants will use the Mumble Melody app undirected daily. Additionally, we will be sending an online platform for participants to conduct at-home testing sessions, in which they will be asked to record their voice during various speech tasks, both with and without the Mumble Melody app.

Participants eligible for this study must:

- (1) Identify as a person who stutters (PWS)
- (2) Be 18 years or older
- (3) Be a US permanent resident
- (4) Have one of the following Apple devices which are compatible with the Mumble Melody application:
  - (a) iPhone with iOS 12.0 or later
  - (b) iPad with iPadOS 12.0 or later
  - (c) iPod touch with iOS 12.0 or later
  - (d) Mac with macOS 11.0 or later and an Apple M1 chip or later
- (5) Have a SEPARATE browser-supporting device with a microphone
- (6) Be able to conduct the study in English
- (7) Qualify based on the initial screening evaluation

Data we will be collecting from participants includes:

- Which modes subjects use each day, and for how long
- Voice recordings for each testing session
- Survey data

Hypotheses that we are testing include:

- 1. Speech fluency will increase significantly from baseline compared to modes within one testing session
- 2. Speech fluency will increase significantly over time (from each session to the next one)

# **Study Flowchart:**

Below is an outline of all steps involved in this study:

### **Protocol Details:**



\*Daily use of the Mumble Melody app between weekly assessments

Each testing session will be laid out as below.

For the Screening Session, a shortened version will be given with no modes and a reading passage will be included.

For the Baseline Testing Session, a quick tutorial on downloading and using the Mumble Melody app will be included.

For the Final Testing Session, a reading passage will be included.

#### **TESTING SESSION #N:**

Home Page:

Welcome to the Week N Testing Session for the Mumble Melody Longitudinal Study on Stuttering

Total Session Time: ~30 MINUTES

About this Session

Here is how the session will take place today:

Step 1: Initial Questions

Step 2: Audio Check

Step 3: Initial voice recording tasks (open-ended questions)

Step 4-7: Voice recording tasks using 4 auditory feedback modes on the Mumble Melody app, which will change the way you hear your voice

Step 8: Final voice recording tasks to share your experience with us

## Materials Needed

- 1) Apple device to use the Mumble Melody app
- 2) Additional browser-supporting device with a microphone (used to conduct this session)
- 3) Wired headphones (shipped to you for the study)
- 4) Lightning-to-headphone jack adapter (shipped to you for the study)

Ready to Get Started?

Click the Join button below:

Join

## Questions (1 min):

TIME REMAINING: ~27 min

Please answer the following questions:

How would you describe your speaking fluency today, compared to your usual fluency?

- My stutter is more severe today
- Same
- My stutter is more mild today

During this step, we will link your submission for this session to your Mumble Melody User ID. In order to do this, please enter the Mumble Melody app on your Apple device and tap the "User ID" button on the home page. The 8-digit ID User ID will be displayed.

| - | Input you | r 8-digit | User ID | below: |
|---|-----------|-----------|---------|--------|
|---|-----------|-----------|---------|--------|

Submit

Click "Next" below: Next

Voice Check (1 min):

TIME REMAINING: ~26 min

For each speaking task, you should click the Record button before speaking and speak for the entire duration. When speaking, try your best to avoid using word replacements or other strategies you typically may use to mask or reduce your stutter. Feel free to stutter freely while speaking.

Before we start, let's test your microphone. Click on the Record button below and say something out loud like "Testing 1, 2, 3". Recording will stop automatically after 5 seconds. Click Play to hear your recording. If you hear background noise, please go to a quieter place and try again by selecting Redo recording. If it sounds good, click Next above.

- Subject Records (5s)

Click "Next" below Next

Testing Session (4 min x 6):

Baseline (no AAF mode), Unaltered, Whisper, Reverb, Harmonize, Final (no AAF mode)

For each speaking task, you should click the Record button before speaking and speak for the entire duration. When speaking, try your best to avoid using word replacements or other strategies you typically may use to mask or reduce your stutter. Feel free to stutter freely while speaking.

We will be asking you a set of open questions. For some questions, you may have the option to select the question you would most like to answer. For each task, record your voice using the Record feature. You will see a countdown and are required to speak for the ENTIRE time of the countdown. If you run out of content towards the prompt, please continue speaking until the countdown ends. Please be aware that researchers will be reviewing these recordings

- I am ready to begin

In this section, we will be testing the mode.

On the device in which you are using Mumble Melody, please:

- (1) Attach your headphones to your Apple device
- (2) Wear your headphones
- (3) Open the Mumble Melody app
- (4) Select the "Modes" button
- (5) Select the "\_\_\_\_" mode
- (6) Test the mode by repeating a few words out loud (for example, "Testing 1, 2, 3") and adjust your volume until you comfortably can hear the mode being used.

If you would like to hear what this mode should sound like, here is a link to our demo beginning at this mode:

When you are able to hear the Mumble Melody mode, click Continue below.

- Continue

Which of the following two questions would you like to answer? Please think about your answer prior to clicking Record, and speak for the ENTIRE duration:

- Question 1: Subject Records (90s)

Which of the following two questions would you like to answer? Please think about your answer prior to clicking Record, and speak for the ENTIRE duration:

- Question 2: Subject Records (90s)

# Submit Responses (1 min):

Thank you for completing the N testing session for this study!

When you are ready, click "Finish" to send us your results. If you have any issues at all, click the "Download" button on the sidebar to export a file with your submission and email us at mumblemelody@mit.edu so we can troubleshoot and get the files sent our way.

Please click "Finish" below to submit your responses. You can additionally click the "Download" button on sidebar if you wish to download a personal copy of your data.

Finish

#### **INITIAL SURVEY:**

The below survey will be provided.

An additional option to take the "Overall Assessment of the Speaker's Experience of Stuttering (OASES™)" will also be provided.

#### Questions:

- 1. What is your age?
- 2. What is your sex at birth?
  - a. Female
  - b. Male
- 3. What is your gender?
  - a. Woman
  - b. Man
  - c. Trans woman
  - d. Trans man
  - e. Non-binary
  - f. Prefer not to disclose
  - g. Other, please specify

| 4 | i. Please specify your gender: |
|---|---|
| 4. | Is English your main spoken language? a. Yes |
| | b. No |
| | <ul> <li>i. What is your main spoken language?</li> <li>ii. What is your proficiency in English?</li> <li>1. Basic: I know vocabulary words and am able to speak simple phrases or sentences, but I have some difficulty understanding native speakers.</li> <li>2. Conversational: I can ask and answer questions and participate in simple conversations on topics.</li> <li>3. Proficient: I am skilled in the language but am at a less-advanced level than a native or fluent speaker.</li> <li>4. Fluent: I have a high level of language proficiency in the language</li> </ul> |
| 5. | Do you stutter? Or have you ever stuttered? |
| | <ul> <li>a. Yes</li> <li>b. No</li> <li>c. Maybe</li> <li>d. Yes in the past but not anymore</li> <li>e. Other, please specify <ul> <li>i. Please specify:</li> </ul> </li> </ul> |
| 6. | Do you currently have any other conditions that may affect speech, voice, or language? |
| | a. No |
| | b. Aphasia |
| | c. Amusia |
| | d. Apraxia |
| | e. Parkinson's disease |
| | f. Any language disorder |
| | g. Any learning disability |
| | h. Dyslexia |
| | i. Attention Deficit Hyperactivity Disorder (ADHD) |
| | j. Other, please specify |
| 7 | <ul><li>i. Please specify:</li><li>If you answered yes to any of the previous conditions, how long have you had them?</li></ul> |
| ١. | a. Since before 2 years old |
| | b. Since 2-5 years old |
| | c. Since 5-7 years old |
| | d. Since 7-10 years old |
| | e. Since 10-18 years old |
| | f. Since after 18 years old |
| | g. I don't know |
| 8. | Have you previously ever had any other conditions that may affect speech, voice, or |
| | language? |
| | a. No |
| | b. Aphasia |
| | c. Amusia |
| | d. Apraxia |
| | e. Parkinson's disease |
| | f. Any lography disability |
| | <ul><li>g. Any learning disability</li><li>h. Dyslexia</li></ul> |
| | n. Dysickia |

| | i. | Attention Deficit Hyperactivity Disorder (ADHD) |
|---|---|---|
| | j. | Other, please specify i. Please specify: |
| a | If you | <ul> <li>i. Please specify:</li> <li>answered yes to any of the previous conditions, how long did you have them?</li> </ul> |
| ٥. | | Starting from before 2 years old |
| | | Starting from 2-5 years old |
| | | Starting from 5-7 years old |
| | | Starting from 7-10 years old |
| | | Starting from 10-18 years old |
| | | Starting from after 18 years old |
| | | I don't know |
| 10. | _ | did you start stuttering? |
| | | Before 2 years old |
| | | 2-5 years old |
| | | 5-7 years old |
| | d. | 7-10 years old |
| | e. | 10-18 years old |
| | f. | After 18 years old |
| | g. | I don't know |
| 11. | | ould you rate your fluency? |
| | | Mild stutter |
| | | Mild/moderate stutter |
| | | Moderate stutter |
| | | Moderate/Severe Stutter |
| | | Severe stutter |
| 12. | | s your education level? |
| | | No schooling completed |
| | | Nursery school to 8th grade |
| | | Some high school, no diploma |
| | | High school graduate, diploma or equivalent (ex: GED) |
| | f. | Some college credit, no degree Trade/technical/vocational training |
| | | Associate's degree |
| | g.<br>h | Bachelor's degree |
| | i. | Master's degree |
| | | Doctorate degree |
| 13 | • | is your household composition? |
| | | Single, never married |
| | | Married or domestic partnership |
| | | Widowed |
| | | Divorced |
| | | Separated |
| 14. | | ou right or left handed? |
| | | Right handed |
| | b. | Left Handed |
| | C. | Ambidextrous |
| | | i. If ambidextrous, what activities do you use each side for? |
| 15. | | you ever been or are you currently going to speech therapy? |
| | | Yes, currently |
| | | Yes, in the past but not anymore |
| | C. | Never |

| | <ul><li>(a/b) Does your therapy focus more on accepting or reducing stuttering?</li><li>Accepting</li><li>Reducing</li></ul> |
|---|---|
| | - Both |
| | - Other, please specify - Please specify: |
| 16. Do you | u stutter in your dreams? |
| - | Never |
| b. | Rarely |
| | Occasionally |
| d. | Often |
| | Always |
| | your inner voice/monologue stutter? |
| | Never |
| | Rarely |
| | Occasionally |
| | Often |
| | Always |
| | ere particular words or sounds for which you stutter more? |
| | are some instances in which you feel you stutter more? |
| | When talking with family |
| | When talking alone |
| | When reading out loud |
| | When talking to children |
| | When talking to pets |
| | When talking with friends |
| | When talking with friends When talking with coworkers |
| i. | In social situations with strangers |
| | —————————————————————————————————————— |
| | During interviews |
| I. | After having a couple of drinks |
| | When talking on the phone |
| | When talking on Zoom or another video call |
| | When talking in front of people |
| p. | When giving a presentation |
| • | Other: |
| • | i. Please specify: |
| 20. What a | are some instances in which you feel you stutter less? |
| a. | When talking with family |
| b. | When talking alone |
| C. | When reading out loud |
| | When talking to children |
| e. | When talking to pets |
| f. | When singing |
| _ | When talking with friends |
| | When talking with coworkers |
| į. | In social situations with strangers |
| j. | When talking to people of authority |
| | During interviews |
| I. | After having a couple of drinks |

| | | When talking on the phone |
|---|---|---|
| | | When talking on Zoom or another video call |
| | | When talking in front of people Other: |
| | ρ. | i. Please specify: |
| 21 | Can vo | ou anticipate that you will stutter a short instant before stuttering? |
| | | Never |
| | | Rarely |
| | | Occasionally |
| | | Often |
| | e. | Always |
| 22. | | ften do you use different words when you think you may stutter? |
| | | Never |
| | | Rarely |
| | | Occasionally |
| | | Often |
| 22 | | Always |
| 23. | | u have any other strategies to compensate for stuttering or to increase fluency? noice of word, slowing down, whispering, preparation, pull-out, preparatory set, |
| | etc.?) | loice of word, slowing down, whispering, preparation, pull-out, preparatory set, |
| 24 | | u try to hide your stuttering? In what ways? |
| | | have relatives who stutter? |
| | - | Yes |
| | | i. If yes, how are you related to them? |
| | b. | No ——— |
| | C. | I don't know |
| 26. | | u sing or play a musical instrument? |
| | | Yes, I sing |
| | b. | Yes, I play a musical instrument |
| | | i. What instrument do you play? |
| | | 1. Piano |
| | | <ol> <li>Recorder</li> <li>Guitar (classic, electric, folk, bass, etc.)</li> </ol> |
| | | 4. Violin |
| | | 5. Percussion/drums |
| | | 6. Other: |
| | | a. Please specify: |
| | C. | Yes, both |
| | d. | No |
| 27. | | nany years of musical training do you have in singing? |
| | | None |
| | | Less than 1 year |
| | | 1-2 years |
| | | 2-5 years |
| | | 5-7 years |
| | | 7-10 years Over 10 years |
| 28 | | nany years of musical training do you have in playing a musical instrument? |
| 20. | | None |
| | | Less than 1 year |
| | | 1-2 years |

| | d. 2-5 years |
|---|---|
| | e. 5-7 years |
| | f. 7-10 years |
| 00 | g. Over 10 years |
| 29 | . How often do you experience verbalized mental thoughts (rehearsing talking in your |
| | head?) |
| | a. All the time |
| | b. A few times an hour |
| | c. A few times a day |
| | d. Less than once a day |
| | e. Never |
| FINIAL | OUDVEW. |
| | . SURVEY: |
| ine be | elow survey will be provided. |
| Questi | ione: |
| | After using it for a month I felt like this app affected my way of speaking/my speech: |
| 1. | a. Negatively |
| | <ul><li>b. Positively</li><li>c. Neutrally (it did change my speech but not in a way that felt good or bad)</li></ul> |
| | <ul><li>d. It didn't affect my speech at all</li><li>e. Other</li></ul> |
| 2 | If it affected your speech, please explain how it did so and why you think this effect is |
| ۷. | positive/negative/neutral: |
| 3 | I feel like this app can make a positive impact on my fluency over a matter of days. |
| ٥. | a. Strongly Disagree |
| | b. Disagree |
| | c. Neutral/Unsure |
| | d. Agree |
| 1 | e. Strongly Agree Please elaborate on why you feel this way: |
| | I feel like this app can make a positive impact on my fluency over a matter of weeks. |
| J. | a. Strongly Disagree |
| | <ul><li>b. Disagree</li><li>c. Neutral/Unsure</li></ul> |
| | 5 5 7 7 |
| 6 | e. Strongly Agree |
| | Please elaborate on why you feel this way: I feel like this app can make a positive impact on my fluency over a matter of months. |
| 7. | a. Strongly Disagree |
| | 0, 0 |
| | <ul><li>b. Disagree</li><li>c. Neutral/Unsure</li></ul> |
| | d. Agree |
| 0 | e. Strongly Agree |
| o.<br>0 | Please elaborate on why you feel this way: |
| 9. | I feel more confident in my speech after using this app for 1 month. |
| | a. Strongly Disagree |
| | b. Disagree |
| | c. Neutral/Unsure |
| | d. Agree |
| | e. Strongly Agree |

| 10. Please elaborate on why you feel this way: 11. This tool in comparison to other assistive technologies that I have used in the past is: a. Much less effective b. Slightly less effective c. About the same d. Slightly more effective e. Much more effective |
|---|
| <ul><li>f. Not applicable</li><li>12. Please describe any other assistive technology that you have used and explain why this</li></ul> |
| tool is more or less helpful: |
| 13. Do you have any comments on the app's interface? |
| 14. Do you have any comments on the app's convenience? |
| 15. Do you have any comments on the app's effect? |
| 16. Do you have any comments on the app's influence on your stutter? |
| <ul><li>17. Do you have any comments on the app's influence on your interactions with others?</li><li>18. Outside of the testing sessions, which situations did you find that you used the app the most?</li></ul> |
| 10. Outside of the testing sessions, which situations did you find that you used the app the most: |
| 19. What situations do you think that the app could be used the most? 20. Which of these situations do you find that the app could be useful for people who stutter? (check |
| all that apply) |
| <ul><li>a. Zoom calls</li><li>b. Conversations while hanging out with friends</li></ul> |
| c. At the workplace in person |
| d. At the workplace virtually |
| e. At home with family |
| f. Speaking by yourself for practice |
| g. Speaking while reading out loud |
| 21. Overall I feel this app made me |
| a. Stutter less |
| b. Stutter more |
| c. Initially made me stutter less and then stopped working |
| <ul> <li>d. Initially made me stutter more and then starting making me stutter less</li> <li>e. Stutter the same amount as I usually do</li> </ul> |
| f. None of the above |
| 22. Please explain further if you would like: |
| 23. Do you think this app could be useful for people who stutter in general? |
| a. Yes |
| b. No |
| c. Maybe |
| 24. Do you think the unaltered mode could be useful for people who stutter in general? |
| a. Yes |
| b. No |
| <ul><li>c. Maybe</li><li>25. Do you think the whisper mode could be useful for people who stutter in general?</li></ul> |
| a. Yes |
| b. No |
| c. Maybe |
| 26. Do you think the reverb mode could be useful for people who stutter in general? |
| a. Yes |
| b. No |
| c. Maybe |

| 27. Do you think the harmonize mode could be useful for people who stutter in general? |
|---|
| a. Yes |
| b. No |
| c. Maybe |
| 28. What features of the app would prevent you from continuing to use it? |
| 29. How could you see this app being used in the future? |
| 30. What barriers do you foresee in others using this app? |
| 31. Mumble Melody is still in early stages of development and we would appreciate any feedback or recommendations. Do you have any suggestions for how we can improve the app? |
| 32. Is there anything else you would like us to know? |